CLINICAL TRIAL: NCT06357780
Title: Closed-loop syncHronization vErsuS convenTional Synchronization in sPontaneously Breathing Adult Nonivasive Ventilation Patients (CHEST-SPAN) - a Randomized Cross-over Trial
Brief Title: Closed-loop syncHronization vErsuS convenTional Synchronization in sPontaneously Breathing Adult Nonivasive ventilationPatients
Acronym: CHESTSPAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 240396837
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Acute Respiratory Failure; Acute Respiratory Distress Syndrome; Chronic Respiratory Failure
Keywords: Acute respiratory failure (ARF); noninvasive ventilation; Closed-loop; synchronization; patient ventilator asynchrony
MeSH Terms: conditions — Respiratory Distress Syndrome; Patient-Ventilator Asynchrony | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Close-loop synchronization controller (Experimental): 30 minutes period where the pressure support of spontaneous effort will be automatically titrated based on pressure and flow waveform analysis obtained from the patient during NIV mode.
  Interventions: Other: close-loop synchronization controller with spontaneous mode
- Conventional (Active Comparator): 30 minutes period where the synchronization of pressure support of patient effort during NIV mode will be manually set.
  Interventions: Other: Conventional

INTERVENTIONS:
Other: close-loop synchronization controller with spontaneous mode — 30 minutes period where the pressure support of spontaneous effort will be automatically titrated based on pressure and flow waveform analysis obtained from the patient during NIV mode.
  Arms: Close-loop synchronization controller
Other: Conventional — 30 minutes period where the synchronization of pressure support of patient effort during NIV mode will be manually set.
  Arms: Conventional

SUMMARY:
The study is a multicentric prospective randomised cross-over study. It evaluates the compatibility of patients with the device without altering the routine treatment applied. During this evaluation, either the clinician-adjusted values on the device or the standard pre-set values are used to obtain hourly and 30-minute PVA (Patient Ventilator Asynchrony) recordings. These recordings will be analysed offline to identify the settings used and to compare the hourly and 30-minute PVA (Patient Ventilator Asynchrony) values when synchronisation is automatically set. The relationships and differences between these values will be analysed. For this purpose, the IntelliSync+ option, already available on the device, will be used. This software continuously analyses waveform signals at least a hundred times per second. This allows for the immediate detection of patient efforts and the initiation of inspiration and expiration in real time, thereby replacing traditional trigger settings for inspiration and expiration. If the patient is already synchronised with this option, it will then be possible to switch to traditional synchronisation settings for comparison. Statistical analyses will be conducted using SPSS 24.0, JASP (Just Another Statistical Programme), Jamovi ( fork of JASP), or R software. Initially, all numerical and categorical data will be evaluated using descriptive statistical methods. The distributions of numerical variables will be examined using visual (histograms and probability plots) and analytical methods (Kolmogorov-Smirnov/Shapiro-Wilk tests). Mean/SD (standard deviation) or median/interquartile range (IQR) will be used as measures of distribution. For comparing numerical data that follows a normal distribution, the Student-t test will be used, and for non-normally distributed data, the Mann-Whitney U or Wilcoxon signed-rank tests will be employed. PVA (Patient Ventilator Asynchrony) values will be statistically compared. For the analysis of categorical data, the Chi-Square test will be applied. Bayesian analysis may also be used as necessary during the writing of the study. The results obtained will be interpreted and reported by the researchers. Results with a "p" value below 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 18 years of age
* Hospitalized at the ICU or emergency department with the intention of treatment with Noninvasive ventilation at least for the upcoming 2 hours with spontaneous breathing activity
* Written informed consent signed and dated by the patient or one relative in case that the patient is unable to consent, after full explanation of the study by the investigator and prior to study participation

Exclusion Criteria:

* Formalized ethical decision to withhold or withdraw life support
* Patient included in another interventional research study under consent
* Patient already enrolled in the present study in a previous episode of respiratory failure
* Pregnant woman
* Patients deemed at high risk for the need of transportation from an intensive care unit or emergency department to another ward, diagnostic unit or any other hospital
* Hemodynamic instability defined as a need of continuous infusion of epinephrine or norepinephrine > 1 mg/h
* Not being able to obtain reference waveforms due to technical or medical problems
* Vulnerable population
* Increase or decrease of ventilatory support either in pressures, fraction of inspired oxygen or mode of ventilation during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Asynchrony Index | 30 minutes
  [(detectable asynchronies )/(total number of breaths + ineffective efforts)]x100

SECONDARY OUTCOMES:
Major Asynchrony index | 30 minutes
  [(major asynchronies)/(total number of breaths + ineffective efforts)]x100
Minor Asynchrony index | 30 minutes
  [(minor asynchronies)/(total number of breaths + ineffective efforts)]x100
Dyspnea Scale | 30 minutes
  Patient subjective dyspnea scale

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Guven, Associate professor, Principal Investigator — Basaksehir Cam Sakura city Hospital, Istanbul
Locations (1):
- Dr.Suat Seren Chest Diseasees Hospital, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Thille AW, Rodriguez P, Cabello B, Lellouche F, Brochard L. Patient-ventilator asynchrony during assisted mechanical ventilation. Intensive Care Med. 2006 Oct;32(10):1515-22. doi: 10.1007/s00134-006-0301-8. Epub 2006 Aug 1. PMID 16896854
- [Background] Longhini F, Bruni A, Garofalo E, Tutino S, Vetrugno L, Navalesi P, De Robertis E, Cammarota G. Monitoring the patient-ventilator asynchrony during non-invasive ventilation. Front Med (Lausanne). 2023 Jan 19;9:1119924. doi: 10.3389/fmed.2022.1119924. eCollection 2022. PMID 36743668
- [Background] Itagaki T, Akimoto Y, Nakano Y, Ueno Y, Ishihara M, Tane N, Tsunano Y, Oto J. Relationships between double cycling and inspiratory effort with diaphragm thickness during the early phase of mechanical ventilation: A prospective observational study. PLoS One. 2022 Aug 17;17(8):e0273173. doi: 10.1371/journal.pone.0273173. eCollection 2022. PMID 35976965
- [Background] Xu Z, Sheng D, Jiao K, Zhang C, Hao J, Ma D. Factors affecting abnormal triggering with non-invasive ventilators: A before-and-after study. Clin Respir J. 2022 Jun;16(6):450-459. doi: 10.1111/crj.13497. Epub 2022 May 31. PMID 35642081
- [Background] Mojoli F, Pozzi M, Orlando A, Bianchi IM, Arisi E, Iotti GA, Braschi A, Brochard L. Timing of inspiratory muscle activity detected from airway pressure and flow during pressure support ventilation: the waveform method. Crit Care. 2022 Jan 30;26(1):32. doi: 10.1186/s13054-022-03895-4. PMID 35094707